CLINICAL TRIAL: NCT00702663
Title: Seroprevalence of Hepatitis B Infection, Effect of Booster Response, and Significance of Anti-HBc Positivity Amongst Taiwanese Young Adults
Brief Title: Seroprevalence of Hepatitis B Infection and Effect of Booster Response Amongst Taiwanese Young Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Fu-Hsiung Su, Far Eastern Memorial Hospital
Other Study IDs: 96035
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Hepatitis B vaccination; booster effect; Taiwan; young adults
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Hepatitis B DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to observe and evaluate initiate serum anti-HBs titers during entrance health examination among undergraduate freshmen in a university who showed a complete 4-dose HBV vaccination in infancy and whose serum status was (1) HBsAg negative and anti-HBc negative and (2) anti-HBc positive alone. For those students whose anti-HBs <10 mIU/ml, additional HBV vaccination boosters were given according to routine governmental suggested schedules. The anamnestic effect then is observed in both groups. The results of this study may contribute to the analysis of the effectiveness of anti-HBV vaccination twenty years after the commencement of the program and the necessity of initiating HBV booster program among Taiwanese young adults.

DETAILED DESCRIPTION:
Hepatitis-B virus infection is endemic in Taiwan with 90% of the adult population having been previously infected with HBV at some stage in their lives, and with approximately 15 - 20% of the general population being carriers of HBV surface antigen at time of writing. In 1984, Taiwan implemented a hepatitis-B vaccination program for high risk newborns. In 1986, the program was extended to all newborns. At the commencement of the program, the HBV carrier rate amongst children was 9.8 percent. Subsequently, from later reports (namely from the 5-, 10-, 15-, 16-,18-, and 20-year post mass HBV vaccination program commencement follow-up studies), the HBV infection and carrier rates would appear to have been declining continuously. However, the long-term efficacy of such vaccination still has remained as one of the main points of interests amongst Taiwan's public-health officials.

Previous researches indicated that hepatitis B surface antibody (HBsAb) acquired from vaccination would decline over time. However, whether the decline of HBsAb implicated loss of protection to hepatitis B infection remained controversial. Reports pertaining to previously immunized healthcare worker (HCW) found that protective HBsAb still persisted in 76% and 52% of HCW after 3 and 13 years respectively. Anamnestic response was also observed, though the study population were limited. Hepatitis B vaccination has been documented to provide protection to HBV infection for at least 15 years for various age groups. Those who were younger than 4 years had the most pronounced decline or protective HBsAb.

Our previous observations have demonstrated that the implementation of the HBV vaccination program since 1984 had reduced the transmission of HBV in Taiwan. However, an increase of prevalence rate of HBV natural infection (anti-HBc positivity) in 1987 cohort, which may suggest the possibility of protection of HBV mass vaccination has gradually decreasing through years. The waning-off of serum anti-HBs level to no protective level among half of our student population has occurred eighteen years after mass vaccination. As a result, the aim of this study is to observe and evaluate initiate serum anti-HBs titers during entrance health examination among undergraduate freshmen in a university who showed a complete 4-dose HBV vaccination in infancy and whose serum status was (1) HBsAg negative and anti-HBc negative and (2) anti-HBc positive alone. For those students whose anti-HBs <10 mIU/ml, additional HBV vaccination boosters were given according to routine governmental suggested schedules. The anamnestic effect then is observed in both groups. The results of this study may contribute to the analysis of the effectiveness of anti-HBV vaccination twenty years after the commencement of the program and the necessity of initiating HBV booster program among Taiwanese young adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-20 years old college new entrants who had complete 4-dose HB vaccination in their infancy

Exclusion Criteria:

* 18-20 years old college new entrants who did not complete a 4-dose HB vaccination in their infancy

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 18-20 year- old freshmen from a private university from northern Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2007-10; Study Completion 2008-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Hsiung Su, BMBS, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Yuan Ze University, Taipei, Taiwan